CLINICAL TRIAL: NCT00025233
Title: A Phase II Trial of Bevacizumab (rhuMAB VEGF) (NSC #704865) in the Treatment of Persistent and Recurrent Squamous Cell Carcinoma of the Cervix (Group A)
Brief Title: Bevacizumab in Treating Patients With Persistent or Recurrent Cancer of the Cervix
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Gynecologic Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02416; NCI-2012-02416 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000068940; GOG-0227C (Other: Gynecologic Oncology Group); GOG-0227C (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2001-10-11; First posted 2003-01-27 (Estimated); Results first posted 2015-06-29 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Cervical Squamous Cell Carcinoma; Recurrent Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Bevacizumab

ARMS (1):
- Treatment (bevacizumab) (Experimental): Patients receive bevacizumab IV over 30-90 minutes on day 1. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: bevacizumab; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is to see if bevacizumab works in treating patients who have persistent or recurrent cancer of the cervix. Monoclonal antibodies, such as bevacizumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or deliver cancer-killing substances to them.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the cytostatic antitumor activity of bevacizumab, in terms of 6-month progression-free survival (PFS), in patients with persistent or recurrent squamous cell carcinoma of the cervix.

II. Determine the nature and degree of toxicity of this drug in these patients. III. Estimate the distribution of PFS and overall survival for patients treated with this drug.

IV. Determine the frequency of clinical response (partial and complete) in patients treated with this drug.

V. Determine the role of age and initial performance status as prognostic factors in patients treated with this drug.

VI. Determine whether biological and imaging markers are associated with clinical efficacy of this drug, such as 6-month PFS, in these patients.

OUTLINE: This is a multicenter study.

Patients receive bevacizumab IV over 30-90 minutes on day 1. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 19-51 patients will be accrued for this study within 11-38 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed persistent or recurrent squamous cell carcinoma (SCC) of the cervix
* Patients must have received at least 1, but no more than 2, prior cytotoxic chemotherapy regimens for advanced, metastatic, or recurrent SCC of the cervix

  * Chemotherapy administered as a radio-sensitizer does not count as 1 regimen
* Documented disease progression
* At least 1 unidimensionally measurable lesion*

  * At least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
* No tumor involving major blood vessels
* No history or physical evidence of CNS disease, including primary or metastatic brain tumor
* Ineligible for a higher priority Gynecological Oncology Group (GOG) protocol (if one exists), including any active GOG phase III protocol for the same patient population
* Performance status - GOG 0-2 (if received 1 prior regimen)
* Performance status - GOG 0-1 (if received 2 prior regimens)
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* No known bleeding disorder or coagulopathy
* No other active bleeding or pathologic condition that would confer a high risk of bleeding
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* SGOT ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN
* INR ≤ 1.5 (or 2-3 for patients on a stable dose of therapeutic warfarin or low molecular weight heparin)
* PTT < 1.2 times control
* Creatinine ≤ 1.5 times ULN
* Creatinine clearance > 60 mL/min
* No proteinuria

  * Urine protein < 1+ on dipstick or < 30 mg/dL
  * Urine protein < 1000 mg by 24-hour urine collection
* No clinically significant cardiovascular disease
* No uncontrolled hypertension
* No myocardial infarction or unstable angina within the past 6 months
* No New York Heart Association grade II-IV congestive heart failure
* No serious cardiac arrhythmia requiring medication
* No grade II or greater peripheral vascular disease
* No history of stroke within the past 5 years
* No greater than grade 1 sensory or motor neuropathy
* No active infection requiring parenteral antibiotics
* No serious nonhealing wound, ulcer, or bone fracture
* No history or physical evidence of seizures not controlled with standard medical therapy
* No known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* No other invasive malignancy within the past 5 years except nonmelanomatous skin cancer
* No significant traumatic injury within the past 4 weeks
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 3 months after completion of study treatment
* No prior bevacizumab
* At least 3 weeks since prior immunologic agents for SCC of the cervix
* See Disease Characteristics
* Recovered from prior chemotherapy
* No prior non-cytotoxic chemotherapy for persistent or recurrent disease
* At least 1 week since prior hormonal therapy for SCC of the cervix
* Concurrent hormone replacement therapy allowed
* See Disease Characteristics
* Recovered from prior radiotherapy
* Recovered from recent prior surgery
* At least 4 weeks since prior major surgical procedure or open biopsy
* At least 1 week since prior placement of vascular access device or core biopsy
* No concurrent major surgical procedure
* At least 3 weeks since other prior therapy for SCC of the cervix
* No prior anticancer therapy that would preclude study therapy
* No concurrent anticoagulants other than those required to maintain the patency of indwelling IV catheters
* No concurrent chronic daily aspirin greater than 325 mg/day or other nonsteroidal anti-inflammatory medications that are known to inhibit platelet function at doses used for chronic inflammatory diseases

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2002-04; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Monk, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on 4/29/2002 and closed to accrual on 11/6/2006 (suspended from 2/7/2005 to 10/30/2005).
Pre-assignment Details: Patients must have persistent or recurrent squamous cell carcinoma of the cervix with documented disease progression. Patients were required to have measurable disease at time of study entry. They were required to have had a prior cytotoxic regimen.
Groups:
- Bevacizumab: Bevacizumab 15 mg/kg IV, every 3 weeks (one cycle) until disease progression or adverse effects prohibit further therapy
Period: Overall Study
Arm/Group | Bevacizumab
Started | 50
Completed | 46
Not Completed | 4
Not completed — Ineligible: wrong cell type | 1
Not completed — Ineligible: wrong primary | 1
Not completed — Ineligible: improper prior treatment | 1
Not completed — Never treated | 1

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients.
Arm/Group | Bevacizumab
Number analyzed (Participants) | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (9.3)
Age, Customized [Number; unit: participants]
  20-29 years | 1
  30-39 years | 11
  40-49 years | 17
  50-59 years | 12
  60-69 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 45
  Canada | 1
Histologic Type [Number; unit: participants]
  Adenosquamous | 3
  Squamous Cell Carcinoma | 43
International Federation of Gynecology and Obstetrics (FIGO) Stage [Number; unit: participants]
  Unspecified | 1
  Recurrent/Persistent | 45

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival Greater Than 6 Months
Description: Whether or not the patient survived progression-free for at least 6 months.
Time Frame: Every other 3-week treatment cycle for 6 months
Population: Eligible and Treated Patients
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 46
percentage of participants | 23.9 [14.0 to 36.5]

2. Primary Outcome: Maximum Severity of Each Adverse Event Per Patient, Graded According to Common Toxicity Criteria Version 2.0
Description: The maximum severity of each adverse event per patient, graded according to Common Toxicity Criteria version 2.0, is reported. Events were restricted to those reported as at least possibly related to study drug.
Time Frame: Every cycle and 30 days after the end of treatment. (average 5 months)
Population: Eligible and treated patients
Measure: Count of Participants; unit: Participants
Groups:
- Grade 0: Number of patients who did not experience the specified AE.
- Grade 1 (CTCAE v 2.0): Number of patients who experienced a grade 1 event using Common Toxicity Criteria version 2.0
- Grade 2 (CTCAE v 2.0): Number of patients who experienced a grade 2 event using Common Toxicity Criteria version 2.0
- Grade 3 (CTCAE v 2.0): Number of patients who experienced a grade 3 event using Common Toxicity Criteria version 2.0
- Grade 4 (CTCAE v 2.0): Number of patients who experienced a grade 4 event using Common Toxicity Criteria version 2.0
- Grade 5 (CTCAE v 2.0): Number of patients who experienced a grade 5 event using Common Toxicity Criteria version 2.0
Arm/Group | Grade 0 | Grade 1 (CTCAE v 2.0) | Grade 2 (CTCAE v 2.0) | Grade 3 (CTCAE v 2.0) | Grade 4 (CTCAE v 2.0) | Grade 5 (CTCAE v 2.0)
Number analyzed (Participants) | 46 | 46 | 46 | 46 | 46 | 46
Participants
  Leukopenia | 39 | 3 | 3 | 1 | 0 | 0
  Thrombocytopenia | 43 | 3 | 0 | 0 | 0 | 0
  Neutropenia | 42 | 2 | 1 | 1 | 0 | 0
  Anemia | 26 | 8 | 10 | 2 | 0 | 0
  Other hematologic | 41 | 1 | 0 | 4 | 0 | 0
  Allergy | 45 | 1 | 0 | 0 | 0 | 0
  Hypertension | 33 | 4 | 2 | 7 | 0 | 0
  Thrombosis Embolism | 41 | 0 | 0 | 4 | 1 | 0
  Other cardiovascular | 34 | 8 | 2 | 2 | 0 | 0
  Coagulation | 43 | 2 | 0 | 1 | 0 | 0
  Constitutional | 22 | 16 | 6 | 2 | 0 | 0
  Dermatologic | 36 | 5 | 5 | 0 | 0 | 0
  Gastrointestinal | 25 | 7 | 10 | 3 | 1 | 0
  Genitourinary/renal | 34 | 6 | 3 | 2 | 1 | 0
  Hemorrhage | 38 | 5 | 2 | 0 | 1 | 0
  Hepatic | 35 | 11 | 0 | 0 | 0 | 0
  Infection | 40 | 0 | 3 | 2 | 0 | 1
  Metabolic | 29 | 16 | 0 | 1 | 0 | 0
  Neuropathy sensory | 41 | 3 | 2 | 0 | 0 | 0
  Other neurologic | 41 | 2 | 3 | 0 | 0 | 0
  Pain | 27 | 8 | 5 | 6 | 0 | 0
  Pulmonary | 38 | 1 | 5 | 2 | 0 | 0

3. Secondary Outcome: Tumor Response
Description: RECIST 1.0 defines complete response as the disappearance of all target lesions and non-target lesions and no evidence of new lesions documented by two disease assessments at least 4 weeks apart. Partial response is defined as at least a 30% decrease in the sum of longest dimensions (LD) of all target measurable lesions taking as reference the baseline sum of LD. There can be no unequivocal progression of non-target lesions and no new lesions. Documentation by two disease assessments at least 4 weeks apart is required. In the case where the ONLY target lesion is a solitary pelvic mass measured by physical exam, which is not radiographically measurable, a 50% decrease in the LD is required. These patients will have their response classified according to the definitions stated above. Complete and partial responses are included in the objective tumor response rate.
Time Frame: Every other cycle during treatment and at the time of treatment discontinuation. (average 5 months)
Population: Eligible and treated patients.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 46
percentage of participants | 10.9 [4.4 to 21.5]

4. Secondary Outcome: Overall Survival
Description: The observed length of life from entry into the study to death or the date of last contact.
Time Frame: From study entry to death or last contact, up to 5 years.
Population: Eligible and treated patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab
Number analyzed (Participants) | 46
months | 7.3 [6.1 to 10.4]

5. Secondary Outcome: Duration of Progression-free Survival
Description: Progression is defined according to RECIST v1.0 as at least a 20% increase in the sum of LD target lesions taking as reference the smallest sum LD recorded since study entry, the appearance of one or more new lesions, death due to disease without prior objective documentation of progression, global deterioration in health status attributable to the disease requiring a change in therapy without objective evidence of progression, or unequivocal progression of existing non-target lesions.
Time Frame: Every other cycle during treatment, then every 3 months for the first 2 years, then every six months for the next three years and then annually for the next 5 years
Population: Eligible and treated patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab
Number analyzed (Participants) | 46
months | 3.40 [2.53 to 4.53]

6. Secondary Outcome: Performance Status
Description: Performance Status 0 = Fully active, able to carry on all pre-disease performance without restriction Performance Status 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of light or sedentary nature, e.g., light housework, office work Performance Status 2 = Ambulatory and capable of all self care but unable to carry out any work activities. Up and about more than 50% of waking hours.
Time Frame: Baseline
Population: Eligible and treated patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 46
Participants
  Performance Status 0 | 22
  Performance Status 1 | 23
  Performance Status 2 | 1

7. Secondary Outcome: Age at Enrollment
Time Frame: Baseline
Population: Eligible and treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 46
Participants
  20-29 years | 1
  30-39 years | 11
  40-49 years | 17
  50-59 years | 12
  60-69 years | 5

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) occurring during treatment and up to 30 days after stopping the study treatment are reported. Also reported are Serious Adverse Events (SAEs) for up to 5 years after stopping study treatment.
Arm/Group | Bevacizumab
Serious Adverse Events (participants affected / at risk) | 27/46
Other Adverse Events (participants affected / at risk) | 46/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab (N=46)
Anemia (Blood and lymphatic system disorders) | 1
Thrombosis Embolism (Cardiac disorders) | 5
Hypertension (Cardiac disorders) | 1
Constitutional Symptoms Other (General disorders) | 4
Fatigue (General disorders) | 2
Abdominal Pain (General disorders) | 2
Pain other (General disorders) | 1
Nail Changes (Skin and subcutaneous tissue disorders) | 1
Diarrhea Without Colostomy (Gastrointestinal disorders) | 1
Melena/Gi Bleeding (Vascular disorders) | 1
Vaginal Bleeding (Vascular disorders) | 2
Infection With Grade 3/4 Neutropenia (Infections and infestations) | 1
Mood Alteration Depression (Nervous system disorders) | 1
Creatinine (Renal and urinary disorders) | 1
Sinus Tachychardia (Cardiac disorders) | 1
Pelvic Pain (General disorders) | 2
Bone Pain (General disorders) | 1
Myalgia (General disorders) | 1
Renal/Gu Other (Renal and urinary disorders) | 2
Ureteral Obstruction (Renal and urinary disorders) | 2
Constipation (Gastrointestinal disorders) | 3
Rectal Bleeding/Hematochezia (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab (N=46)
Allergic Rhinitis (Immune system disorders) | 5
Allergic Reaction (Immune system disorders) | 1
Inner Ear/Hearing (Ear and labyrinth disorders) | 2
Middle Ear/Hearing (Ear and labyrinth disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 5
Lymphopenia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 10
Transfusion Prbc's (Blood and lymphatic system disorders) | 12
Anemia (Blood and lymphatic system disorders) | 33
Transfusion Platelets (Blood and lymphatic system disorders) | 1
Lymphatics Other (Blood and lymphatic system disorders) | 1
Cardiac Left Ventricular Function (Cardiac disorders) | 1
Sinus Tachycardia (Cardiac disorders) | 4
Arrhythmia Nodal/Junctional Dysrhythmia (Cardiac disorders) | 1
Edema (Cardiac disorders) | 11
Thrombosis Embolism (Cardiac disorders) | 6
Hypertension (Cardiac disorders) | 15
Palpitations (Cardiac disorders) | 2
Prothrombin Time (Vascular disorders) | 1
Coagulation Other (Vascular disorders) | 1
Partial Thromboplastin Time (Vascular disorders) | 5
Rectal Bleeding/Hematochezia (Vascular disorders) | 5
Epistaxis (Vascular disorders) | 1
Vaginal Bleeding (Vascular disorders) | 10
Hematuria No Vaginal Bleeding (Vascular disorders) | 4
Hemoptysis (Vascular disorders) | 1
Fever(No Neutropenia) (General disorders) | 4
Weight Loss (General disorders) | 8
Rigors Chills (General disorders) | 3
Constitutional Symptoms Other (General disorders) | 2
Sweating (General disorders) | 2
Fatigue (General disorders) | 34
Abdominal Pain (General disorders) | 21
Pain Other (General disorders) | 19
Pain Tumor (General disorders) | 5
Neuropathic Pain (General disorders) | 3
Earache (General disorders) | 1
Dyspareunia (General disorders) | 1
Headache (General disorders) | 8
Pelvic Pain (General disorders) | 11
Chest Pain (General disorders) | 6
Bone Pain (General disorders) | 5
Arthralgia (General disorders) | 12
Myalgia (General disorders) | 10
Pain Rectal/Perirectal (General disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 11
Rash Desquamation (Skin and subcutaneous tissue disorders) | 9
Skin Other (Skin and subcutaneous tissue disorders) | 1
Nail Changes (Skin and subcutaneous tissue disorders) | 3
Wound Not-Infectious (Skin and subcutaneous tissue disorders) | 2
Pigmentation Changes (Skin and subcutaneous tissue disorders) | 1
Wound Infectious (Skin and subcutaneous tissue disorders) | 1
Bruising (Skin and subcutaneous tissue disorders) | 3
Dry Skin (Skin and subcutaneous tissue disorders) | 3
Hot Flashes/Flushes (Endocrine disorders) | 6
Anorexia (Gastrointestinal disorders) | 19
Flatulence (Gastrointestinal disorders) | 1
Fistula Intestinal (Gastrointestinal disorders) | 1
Mouth Dryness (Gastrointestinal disorders) | 1
Proctitis (Gastrointestinal disorders) | 2
Dyspepsia/Heartburn (Gastrointestinal disorders) | 3
Fistula Rectal/Anal (Gastrointestinal disorders) | 3
Taste Disturbance (Gastrointestinal disorders) | 2
Diarrhea Without Colostomy (Gastrointestinal disorders) | 9
Constipation (Gastrointestinal disorders) | 21
Stomatitis/Pharyngitis (Gastrointestinal disorders) | 8
Dehydration (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 12
Nausea (Gastrointestinal disorders) | 19
Gi Other (Gastrointestinal disorders) | 4
Hypoalbuminemia (Hepatobiliary disorders) | 9
Sgot(Alt) (Hepatobiliary disorders) | 5
Sgot(Ast) (Hepatobiliary disorders) | 9
Alkaline Phosphatase (Hepatobiliary disorders) | 13
Bilirubin (Hepatobiliary disorders) | 1
Infection No Anc (Infections and infestations) | 1
Infection Without Neutropenia (Infections and infestations) | 17
Hypophosphatemia (Metabolism and nutrition disorders) | 4
Metabolic Other (Metabolism and nutrition disorders) | 11
Hyponatremia (Metabolism and nutrition disorders) | 15
Bicarbonate (Metabolism and nutrition disorders) | 3
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 4
Hypermagnesemia (Metabolism and nutrition disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 19
Hypoglycemia (Metabolism and nutrition disorders) | 6
Hypokalemia (Metabolism and nutrition disorders) | 9
Hypercalcemia (Metabolism and nutrition disorders) | 3
Hypomagnesmia (Metabolism and nutrition disorders) | 11
Muscle Weakness (Metabolism and nutrition disorders) | 2
Tremor (Musculoskeletal and connective tissue disorders) | 1
Speech Impairment (Musculoskeletal and connective tissue disorders) | 1
Hallucinations (Musculoskeletal and connective tissue disorders) | 1
Extrapyramidal (Musculoskeletal and connective tissue disorders) | 2
Depressed Level Of Consciousness (Musculoskeletal and connective tissue disorders) | 1
Confusion (Musculoskeletal and connective tissue disorders) | 1
Mood Alteration Anxiety/Agitation (Musculoskeletal and connective tissue disorders) | 1
Memory Loss (Musculoskeletal and connective tissue disorders) | 1
Insomnia (Musculoskeletal and connective tissue disorders) | 5
Dizziness (Musculoskeletal and connective tissue disorders) | 5
Mood Alteration Depression (Musculoskeletal and connective tissue disorders) | 8
Neuropathy Sensor (Musculoskeletal and connective tissue disorders) | 16
Neuropathy Motor (Musculoskeletal and connective tissue disorders) | 1
Ocular Other (Eye disorders) | 1
Tearing (Eye disorders) | 1
Keratitis (Eye disorders) | 1
Conjunctivitis (Eye disorders) | 1
Vision Flashing Lights/Floaters (Eye disorders) | 1
Double Vision (Eye disorders) | 2
Voice Changes/Stridor/Larynx (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 14
Urinary Frequency/Urgency (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 3
Creatinine (Renal and urinary disorders) | 11
Renal/Gu Other (Renal and urinary disorders) | 3
Urinary Retention (Renal and urinary disorders) | 3
Ureteral Obstruction (Renal and urinary disorders) | 3
Incontinence (Renal and urinary disorders) | 4
Hemoglobinuria (Renal and urinary disorders) | 2
Fistula (Renal and urinary disorders) | 1
Bladder Spasms (Renal and urinary disorders) | 3
Proteinuria (Renal and urinary disorders) | 10
Libido (Reproductive system and breast disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less